CLINICAL TRIAL: NCT07001852
Title: EnDOvascular Therapy for Late WiNdow IschEmic Stroke Patients Selected bY AutoMatic Plain ComputErized Tomography
Acronym: DONE SYMPLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Santiago Ortega Gutierrez (Other)
Collaborators: Fundació Ictus (Unknown)
Responsible Party: Sponsor-Investigator, Santiago Ortega Gutierrez, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202312563
Record Dates: First submitted 2025-05-15; First posted 2025-06-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Stroke Acute
Keywords: large vessel occlusion; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: The DONE SYMPLE Trial follows a parallel assignment model, in which eligible participants are randomly assigned in a 1:1 ratio to one of two study arms: (1) standard medical therapy alone (control group), or (2) standard medical therapy plus endovascular thrombectomy (intervention group). Participants remain in their assigned group for the duration of the study, and outcomes are assessed at predefined time points. This design allows for direct comparison between the intervention and control arms to evaluate the safety and efficacy of endovascular treatment initiated between 6 and 72 hours from last known well, based on selection by non-contrast CT analyzed with automated software.
Who Masked: Outcomes Assessor
Masking Description: Data Analysts: Individuals analyzing the data may also be blinded to the treatment assignment to avoid bias in data interpretation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Therapy + Standard Medical Management (Active Comparator): Participants in this arm will receive standard medical management for acute ischemic stroke plus endovascular therapy (mechanical thrombectomy). Treatment is initiated within 6 to 72 hours of stroke onset and is guided by automated non-contrast CT selection software.
  Interventions: Other: Endovascular Therapy (Mechanical Thrombectomy); Other: Standard Medical Management
- Standard Medical Management Alone (Active Comparator): Participants in this arm will receive standard medical management for acute ischemic stroke without undergoing endovascular therapy. Treatment decisions are made according to institutional protocols and exclude mechanical thrombectomy.
  Interventions: Other: Standard Medical Management

INTERVENTIONS:
Other: Endovascular Therapy (Mechanical Thrombectomy) — Endovascular therapy performed with CE-approved thrombectomy devices, initiated within 6 to 72 hours after stroke onset in patients with anterior circulation large vessel occlusion. The procedure is guided by an automated non-contrast CT detection tool and follows standard device-specific instructions for use.
  Arms: Endovascular Therapy + Standard Medical Management
Other: Standard Medical Management — Standard medical management including therapies such as antiplatelet agents, anticoagulants, blood pressure control, and general supportive care. Delivered in accordance with institutional guidelines for acute ischemic stroke.

SUMMARY:
The DONE SYMPLE Investigator-initiated phase III prospective, randomized, open-label, blinded endpoint-controlled clinical trial.

This clinical trial is a global clinical study testing whether a procedure called endovascular therapy, which removes blood clots from blocked brain arteries, can safely benefit more stroke patients when used up to 72 hours after symptoms begin. Endovacular Therapy is already proven to improve recovery in patients treated within 6 hours, but only when advanced imaging like Computed Tomography (CT) perfusion or Magnetic Resonance Imaging (MRI) is available to guide treatment. Unfortunately, many hospitals, specially in underserved areas, do not have access to this type of imaging.

This trial will investigate whether a basic brain scan called non-contrast CT, which is widely available in hospitals around the world, can be used instead. Special software will automatically analyze the CT scan to help doctors decide if a patient has enough brain tissue left to save with Endovascular Therapy. If this simpler approach works, it could expand access to lifesaving stroke care for more people globally.

The study will enroll 500 adult stroke patients, ages 18 to 80, with a large vessel blockage in the brain's anterior circulation, moderate to severe stroke symptoms, and who are between 6 and 72 hours from when they were last known to be well. All participants will undergo CT imaging analyzed by the automated software. If the scan shows a small core of already damaged brain tissue and a larger area of threatened but still viable brain, the patient will qualify.

Participants will be randomly assigned to receive either standard medical therapy alone or medical therapy plus Endovasculat Therapy which involves inserting a catheter through a blood vessel to reach the brain and using a device to remove the clot. This procedure is performed by trained stroke or neurointerventional specialists. The study is "open-label," meaning patients and doctors know which treatment is given, but the assessment of patient recovery will be done by independent reviewers who do not know the group assignments.

The primary goal is to determine if patients who receive Endovascular Therapy have better recovery at 90 days, measured by a scale called the modified Rankin Scale, which assesses how much disability a patient has after a stroke. The trial will also look at safety (especially brain bleeding after treatment), size and growth of brain injury on follow-up scans, recovery of strength and language, and overall quality of life and survival. Imaging will be reviewed centrally by a specialized team, and results will be analyzed to see how well Endovascular Therapy performs using this new patient selection method.

The DONE SYMPLE Trial is sponsored by Foundacio Ictus in Barcelona Spain and the University of Iowa is the Central Coordinating Center for the Study. It will take place at up to 20 hospitals worldwide. All patients will be followed closely with exams and imaging at specific time points up to 90 days after treatment.

If successful, this trial could change stroke care around the world by proving that Endovascular Therapy can be used safely and effectively even without advanced imaging, using tools available in most hospitals. This could help more stroke patients, especially in rural or resource-limited areas, access treatments that may improve their chances of recovery and reduce long-term disability.

DETAILED DESCRIPTION:
The DONE SYMPLE Trial is a Phase III, multicenter, prospective, randomized, open-label trial with blinded endpoint assessment (PROBE design), evaluating the safety and efficacy of endovascular therapy (EVT) in patients with acute ischemic stroke (AIS) due to anterior circulation large vessel occlusion (LVO) treated between 6 to 72 hours from last known well. The key innovation is the use of non-contrast computed tomography (NCCT) with automated software analysis as the sole selection modality, replacing advanced imaging requirements such as CT perfusion or MRI diffusion-perfusion mismatch.

The trial addresses critical gaps in access to reperfusion therapy by enabling stroke triage and selection using standard NCCT imaging combined with artificial intelligence tools, thereby facilitating inclusion of centers without advanced imaging infrastructure. The selection criteria are based on automated estimation of ischemic core volume (≤70 cc) and evidence of LVO detection, derived from FDA-cleared deep learning algorithms and structured image analysis (e.g., ASPECTS quantification and vessel segmentation).

A total of 500 patients will be randomized 1:1 to either (1) standard medical therapy or (2) EVT plus standard medical therapy. Randomization will be stratified by baseline stroke severity (NIH Stroke Scale), time from symptom onset, core infarct volume, and enrolling site. EVT will be performed using CE-marked or FDA-cleared thrombectomy devices following standard institutional practice.

The primary endpoint is global disability at 90 days, assessed using the utility-weighted modified Rankin Scale (dw-mRS). Secondary efficacy analyses include mRS ordinal shift, dichotomized mRS (0-2), NIHSS change, and angiographic endpoints such as reperfusion success (TICI ≥2b) and first-pass effect (TICI 2c-3 on first attempt). Safety outcomes include symptomatic intracranial hemorrhage (sICH) per Heidelberg criteria, infarct growth on serial imaging, and all-cause mortality.

The statistical framework employs a Bayesian Gaussian model stratified by time-to-treatment intervals (6-24, 24-48, and 48-72 hours). The adaptive enrichment design enables interim analyses after enrollment milestones (n=200, 275, 350, 425) to evaluate futility, efficacy, or harm. The final sample size accounts for 10% potential LVO detection misclassification by automated software and 5% anticipated loss to follow-up.

Imaging is adjudicated centrally by a blinded core laboratory, ensuring uniform quantification of infarct volume and recanalization metrics. Functional outcomes are assessed by trained evaluators blinded to treatment allocation. Trial conduct is overseen by an independent data monitoring committee and a clinical events committee to adjudicate adverse events and outcomes.

By leveraging accessible imaging with automated tools, the DONE SYMPLE Trial aims to demonstrate that safe and effective EVT can be extended to patients beyond 24 hours and in settings without advanced imaging. If positive, the findings will inform future guideline updates and support broader implementation of thrombectomy in underserved populations globally.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age:

   1. Pre-stroke score (mRS) of 0-1 in participants aged 18 to 70 years.
   2. Pre-stroke Modified Rankin Scale (mRS) score of 0 in participants older than 70 years.
2. Presenting with signs and symptoms consistent with an acute ischemic stroke within 24-72 hours from last known well. *
3. Baseline NIHSS ≥8.
4. NCCT imaging indicating the existence of an anterior circulation LVO by an automated software, or CTA (when available).
5. Core volume ≤ 70 cc determined by a deep learning algorithm in automated software and/or ASPECTS scoring ≥ 6. **
6. Arterial puncture within 72 hours (after the first symptoms or LKW).
7. Arterial puncture within 90 minutes from initial CT.
8. Ability to randomize within 72 hours after stroke onset (last seen well).
9. Ability to obtain signed informed consent or subject's Legally Authorized representative (LAR) has signed Consent form ***

   * Patients in the 6-24-hour after Last Known Well (LKW) may be enrolled only in centers where thrombectomy is not offered as standard of care due to the absence of advanced imaging capabilities.

     * In cases of discrepancy between the automated tool LVO detection and volume, and ASPECT Score or CTA judgment or Computed Tomography Angiography CTA findings, ASPECTS and CTA will take precedence.

       * If approved by local ethics committee and country regulations, the investigator is allowed to enroll a patient utilizing emergency informed consent procedures if neither the patient nor the representative or person of trust is available to sign the informed consent form. However, as soon as possible, the patient is informed, and his/her consent is requested for the possible continuation of this research.

Exclusion Criteria:

1. Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test.
2. Known severe allergy (more than a rash) to contrast media uncontrolled by medications.
3. Refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg) despite medication.
4. CT evidence of the following conditions:

   * Midline shift or herniation.
   * Evidence of intracranial hemorrhage.
   * Mass effect with effacement of the ventricles.
5. Bilateral strokes.
6. Clot retrieval previously attempted <6 hours.
7. Treated with thrombolytics >4.5 hours after last seen well.
8. Intracranial tumors.
9. Life expectancy less than 90 days prior to stroke onset.
10. Participation in another randomized clinical trial that could confound the evaluation of the study.
11. Presumed septic embolus, or suspicion of bacterial endocarditis.
12. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept).
13. Any other condition (in the opinion of the site investigator) that precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was performed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Global Disability at 90 Days | 90 days (±14 days)
  Global disability will be measured using the disability-weighted modified Rankin Scale (dw-mRS) at 90 days (±14 days) post-stroke. The dw-mRS is a validated tool that captures the severity of post-stroke disability across seven levels, ranging from no symptoms (0) to death (6). This outcome evaluates whether endovascular therapy (EVT) plus medical management results in superior functional outcomes compared to medical management alone in patients with anterior circulation large vessel occlusion (LVO) strokes treated between 6-72 hours after stroke onset and selected exclusively by automated non-contrast CT imaging.

SECONDARY OUTCOMES:
Ordinal Distribution of the Modified Rankin Scale (mRS) at 90 Days | 90 days (±14 days)
  Global disability will be assessed using the full ordinal distribution of the Modified Rankin Scale (mRS), a 7-point scale that measures functional independence and global disability after stroke. The scale ranges from 0 to 6, where 0 indicates no symptoms and 6 indicates death. Higher scores represent worse outcomes. For the purposes of this analysis, categories 5 (severe disability) and 6 (death) will be collapsed into a single category to enhance statistical robustness.
Proportion of Participants with Functional Independence (mRS 0-2) at 90 Days | 90 days (±14 days)
  Functional independence will be defined as achieving a score of 0 to 2 on the Modified Rankin Scale (mRS), a 7-point scale used to measure the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with higher scores indicating worse outcomes. Scores of 0 to 2 reflect no symptoms, slight disability, or moderate disability with preserved independence.
Change in NIH Stroke Scale (NIHSS) Score at 24 Hours | 24 hours (±16 hours)
  Absolute change in the National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours post-randomization. The NIHSS is a 42-point clinical scale used to assess neurological impairment in patients with stroke. Scores range from 0 to 42, with higher scores indicating greater stroke severity and worse neurological function. A decrease in NIHSS score represents clinical improvement.
Change in NIHSS Score at Day 5 or Discharge | 5 days (±1 day) or at discharge
  Absolute change in the National Institutes of Health Stroke Scale (NIHSS) score from baseline to Day 5 (±1 day) post-randomization or hospital discharge, whichever occurs first. The NIHSS is a validated clinical scale ranging from 0 (no neurological deficit) to 42 (most severe deficit), with higher scores indicating more severe stroke-related impairment. A reduction in score reflects neurological improvement.
Major Early Neurological Improvement at 24 Hours | 24 hours (±16 hours)
  Proportion of participants achieving either a ≥10-point reduction in NIHSS or an NIHSS score of 0-1 at 24 hours. This is a robust early marker of favorable prognosis.
Early Neurological Recovery at 24 Hours | 24 hours (±16 hours)
  Proportion of participants demonstrating early neurological improvement, defined as a ≥4-point reduction in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours post-randomization. The NIHSS is a standardized 42-point scale used to quantify neurological impairment following stroke, where scores range from 0 (no deficit) to 42 (maximum deficit). Higher scores indicate more severe impairment; thus, a decrease of 4 or more points reflects meaningful early neurological
Successful Angiographic Reperfusion | At the end of the endovascular procedure
  Defined as achieving modified Thrombolysis in Cerebral Infarction (mTICI) grade ≥2b at the end of the endovascular procedure, indicating adequate perfusion of the downstream territory.
First Pass Recanalization Rate | Perioperative/Periprocedural
  Proportion of patients achieving mTICI 2c or 3 on the first pass of the thrombectomy device in the intervention arm, a strong predictor of improved outcomes.
Workflow Efficiency Metrics | From hospital arrival to procedure completion
  Quantitative time intervals including: door-to-CT, CT-to-arterial puncture, puncture-to-reperfusion, and puncture-to-final angiogram, used to assess procedural timeliness.
Length of Inpatient Stay | From hospital admission to discharge (up to 90 days post-randomization)
  Total number of days from admission to discharge from the index hospitalization.
Discharge Disposition | At hospital discharge (up to 90 days post-randomization)
  Classification of discharge destination as home, acute rehabilitation, skilled nursing facility, long-term care, or other.
Health-Related Quality of Life (HRQoL) at 90 Days | 90 days (±14 days)
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument, a validated patient-reported outcome measure that evaluates five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 5-point scale (1 = no problems; 5 = extreme problems). Responses are used to generate an index value ranging from less than 0 (states worse than death) to 1 (full health), with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tudor Jovin, MD, Principal Investigator — Cooper University Health Care; Marc Ribo, MD, Principal Investigator — Hospital Vall d"Hebron Barcelona
Locations (2):
- University of Iowa, Iowa City, Iowa, United States
- Erebouni Medical Center, Yerevan, Armenia

REFERENCES:
- [Background] Jovin TG, Nogueira RG, Lansberg MG, Demchuk AM, Martins SO, Mocco J, Ribo M, Jadhav AP, Ortega-Gutierrez S, Hill MD, Lima FO, Haussen DC, Brown S, Goyal M, Siddiqui AH, Heit JJ, Menon BK, Kemp S, Budzik R, Urra X, Marks MP, Costalat V, Liebeskind DS, Albers GW. Thrombectomy for anterior circulation stroke beyond 6 h from time last known well (AURORA): a systematic review and individual patient data meta-analysis. Lancet. 2022 Jan 15;399(10321):249-258. doi: 10.1016/S0140-6736(21)01341-6. Epub 2021 Nov 11. PMID 34774198
- [Background] Desai SM, Haussen DC, Aghaebrahim A, Al-Bayati AR, Santos R, Nogueira RG, Jovin TG, Jadhav AP. Thrombectomy 24 hours after stroke: beyond DAWN. J Neurointerv Surg. 2018 Nov;10(11):1039-1042. doi: 10.1136/neurintsurg-2018-013923. Epub 2018 May 28. PMID 29807887
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510